CLINICAL TRIAL: NCT01077115
Title: Extent of Surgical Trauma in Open and Laparoscopic Cholecystectomy
Acronym: ESTOLC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Montenegro (Other Government)
Collaborators: Medical School of Podgorica, Montenegro (Unknown); General Hospital Berane, Montenegro (Unknown)
Responsible Party: Dr Miodrag Radunovic, MD, PhD, Ministry of Health, Montenegro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOHMNE001
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2010-02

CONDITIONS: Chronic Calculous Cholecystitis
Keywords: Cholecystectomy; Cholecystitis; Laparoscopy; Cholelithiasis; Operative trauma
MeSH Terms: conditions — Cholecystitis; Cholelithiasis | interventions — Cholecystectomy, Laparoscopic; Conversion to Open Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic cholecystectomy (Experimental)
  Interventions: Procedure: Laparoscopic cholecystectomy
- Open cholecystectomy (Active Comparator)
  Interventions: Procedure: Open Surgery

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy
  Arms: Laparoscopic cholecystectomy
Procedure: Open Surgery
  Arms: Open cholecystectomy

SUMMARY:
The aim of this work is to evaluate which of the two types of operation (traditional/open and laparoscopic) has more impact on patients who were operated electively due to their chronic calculous cholecystitis.

DETAILED DESCRIPTION:
The prospective, single center, randomized study includes 120 patients who are operated electively - 60 patients operated laparoscopically and 60 patients operated traditionally. Biohumoral and endocrine parameters of response to trauma are determined from 24 hour urine and blood: adrenalin, noradrenalin, metabolites of corticosteroid hormone - 17- hydroxyl and 17- keto steroid (HPLC method), C reactive protein and albumin, glycemia, creatine phosphokinase, lactate dehydrogenase, sedimentation of erythrocytes and serum concentration of potassium.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Calculous Cholecystitis

Exclusion Criteria:

* Previous Biliary Surgery
* Cholangitis
* Obstructive jaundice

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2003-06; Primary Completion 2004-06 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
To determine biohumoral and endocrine parameters of response to trauma | first 24h after the surgical intervention
  Urine and blood biochemical analyses: adrenalin, noradrenalin, metabolites of corticosteroid hormone - 17- hydroxyl and 17- keto steroid (HPLC method), C reactive protein and albumin, glycemia, creatine phosphokinase, lactate dehydrogenase, sedimentation of erythrocytes and serum concentration of potassium

CONTACTS AND LOCATIONS:
Overall Officials: Miodrag Radunovic, MD, PhD, Principal Investigator — Ministry of Health, Republic of Montenegro
Locations (1):
- Ministry of Health, Podgorica, Montenegro

REFERENCES:
- [Background] Donald RA, Perry EG, Wittert GA, Chapman M, Livesey JH, Ellis MJ, Evans MJ, Yandle T, Espiner EA. The plasma ACTH, AVP, CRH and catecholamine responses to conventional and laparoscopic cholecystectomy. Clin Endocrinol (Oxf). 1993 Jun;38(6):609-15. doi: 10.1111/j.1365-2265.1993.tb02142.x. PMID 8392916
- [Background] Crema E, Ribeiro EN, Hial AM, Alves Junior JT, Pastore R, Silva AA. Evaluation of the response of cortisol, corticotropin and blood platelets kinetics after laparoscopic and open cholecystectomy. Acta Cir Bras. 2005 Sep-Oct;20(5):364-7. doi: 10.1590/s0102-86502005000500005. Epub 2005 Sep 5. PMID 16186960
- [Background] Mrksic M, Cabafi Z, Feher I, Mirkovic M. [Surgical trauma in laparoscopic and classical cholecystectomy]. Med Pregl. 2001 Jul-Aug;54(7-8):327-31. Croatian. PMID 11905180
- [Background] Bisgaard T, Rosenberg J, Kehlet H. From acute to chronic pain after laparoscopic cholecystectomy: a prospective follow-up analysis. Scand J Gastroenterol. 2005 Nov;40(11):1358-64. doi: 10.1080/00365520510023675. PMID 16334446
- [Background] Ros A, Nilsson E. Abdominal pain and patient overall and cosmetic satisfaction one year after cholecystectomy: outcome of a randomized trial comparing laparoscopic and minilaparotomy cholecystectomy. Scand J Gastroenterol. 2004 Aug;39(8):773-7. doi: 10.1080/00365520410005540. PMID 15513364
- [Background] Schirmer BD, Winters KL, Edlich RF. Cholelithiasis and cholecystitis. J Long Term Eff Med Implants. 2005;15(3):329-38. doi: 10.1615/jlongtermeffmedimplants.v15.i3.90. PMID 16022643
- [Background] Chen L, Tao SF, Xu Y, Fang F, Peng SY. Patients' quality of life after laparoscopic or open cholecystectomy. J Zhejiang Univ Sci B. 2005 Jul;6(7):678-81. doi: 10.1631/jzus.2005.B0678. PMID 15973772
- [Background] Nilsson E, Ros A, Rahmqvist M, Backman K, Carlsson P. Cholecystectomy: costs and health-related quality of life: a comparison of two techniques. Int J Qual Health Care. 2004 Dec;16(6):473-82. doi: 10.1093/intqhc/mzh077. PMID 15557357
- [Background] Agnifili A, Ibi I, Guadagni S, Verzaro R, Gianfelice F, Mancini E, De Bernardinis G, Silvi B, Leonardis F. [Perioperative pain and stress: a comparison between video laparoscopic cholecystectomy and "open" cholecystectomy]. G Chir. 1993 Sep;14(7):344-8. Italian. PMID 8286176
- [Background] Hakanson E, Rutberg H, Jorfeldt L, Wiklund L. Endocrine and metabolic responses after standardized moderate surgical trauma: influence of age and sex. Clin Physiol. 1984 Dec;4(6):461-73. doi: 10.1111/j.1475-097x.1984.tb00132.x. PMID 6542833
- [Background] Mealy K, Gallagher H, Barry M, Lennon F, Traynor O, Hyland J. Physiological and metabolic responses to open and laparoscopic cholecystectomy. Br J Surg. 1992 Oct;79(10):1061-4. doi: 10.1002/bjs.1800791024. PMID 1422720
- [Background] Kiviluoto T, Siren J, Luukkonen P, Kivilaakso E. Randomised trial of laparoscopic versus open cholecystectomy for acute and gangrenous cholecystitis. Lancet. 1998 Jan 31;351(9099):321-5. doi: 10.1016/S0140-6736(97)08447-X. PMID 9652612
- [Background] Johansson M, Thune A, Nelvin L, Lundell L. Randomized clinical trial of day-care versus overnight-stay laparoscopic cholecystectomy. Br J Surg. 2006 Jan;93(1):40-5. doi: 10.1002/bjs.5241. PMID 16329083
- [Background] Udelsman R, Chrousos GP. Hormonal responses to surgical stress. Adv Exp Med Biol. 1988;245:265-72. doi: 10.1007/978-1-4899-2064-5_21. PMID 2852458
- [Background] Baxter JN, O'Dwyer PJ. Pathophysiology of laparoscopy. Br J Surg. 1995 Jan;82(1):1-2. doi: 10.1002/bjs.1800820102. No abstract available. PMID 7881922